CLINICAL TRIAL: NCT06305468
Title: Prognosis of Disseminated and Cerebral Toxoplasmosis Hospitalized in Intensive Care in the Era of PCR Diagnosis - Toxoplasmosis in ICU (TOXIC)
Brief Title: Prognosis of Disseminated and Cerebral Toxoplasmosis Hospitalized in Intensive Care in the Era of PCR Diagnosis
Acronym: TOXIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240055
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Toxoplasmosis
Keywords: toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Toxoplasmosis is a common infection whose clinical severity can sometimes justify admission to intensive care, especially in immunocompromised patients.

This study should make it possible to evaluate the impact of different anti-infective treatment regimens and to highlight clinical-biological and prognostic differences depending on the type of underlying immunosuppression.

DETAILED DESCRIPTION:
Toxoplasmosis is a common infection whose clinical severity can sometimes justify admission to intensive care, especially in immunocompromised patients. There are different clinical forms: cerebral toxoplasmosis on the one hand, and disseminated form on the other. However, few studies have looked at the prognosis of severe toxoplasmosis hospitalized in intensive care. Historically, the diagnosis was made according to a set of clinical-biological arguments and the response to the test treatment. Polymerase chain reaction (PCR) diagnosis has significantly changed diagnostic management. One study reported 38 cases of disseminated toxoplasmosis (positive blood PCR or Bronchoalveolar lavage (BAL) or bone marrow or parasite found on biopsy of at least one organ) in HIV-infected patients who received allogeneic transplants over a 10-year period (2002 to 2012).

This study did not include an analysis of these 2 subgroups, which probably have their own specificity, and no comparison of the efficacy of the different treatment regimens was performed. Another study reported 100 cases of cerebral toxoplasmosis in HIV patients hospitalized in intensive care units; only 21% of cases had a positive PCR on cerebrospinal fluid (CSF). The standard curative treatment for toxoplasmosis is pyrimethamine-sulfadiazine per os. However, in intensive care, trimethoprim-sulfamethoxazole (TMP-SMX) IV or the combination of oral pyrimethamine and IV clindamycin are sometimes used if the parenteral route is preferred. No studies have been carried out in intensive care. The latest U.S. recommendations report that "some specialists will use TMP-SMX IV (IB) or oral pyrimethamine plus IV clindamycin (IIIC) as initial treatment in severe patients requiring parenteral therapy."

This descriptive study focuses on a particularly severe opportunistic infection of the immunocompromised and should allow to better specify the clinico-biological presentation of patients with disseminated or cerebral toxoplasmosis, in particular according to the type of underlying immunosuppression, in order to allow early detection of this severe complication. The identification of new categories of patients at risk, prognostic factors and the study of the impact of the use of different treatment regimens could make it possible to improve its management in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in intensive care
* At least 1 organ failure (SOFA> or =2)
* PCR toxoplasmosis on CSF, blood, BAL, or bone marrow positive within 7 days before or after admission to ICU

Exclusion Criteria:

* Post-mortem diagnosis
* Primary outcome not available
* Patient living informed and not opposed to the reuse of their data in this research.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care for toxoplasmosis (positive toxoplasmosis PCR) between 2012 (01/01/2012) and 2023 (02/01/2023)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate in intensive care. | 11 years
  The aim is to determine the impact of the anti-infective treatment regimen used on the prognosis of patients with severe toxoplasmosis in intensive care.

SECONDARY OUTCOMES:
Hospital mortality rate | 11 years
Length of stay in intensive care | 11 years
Duration of mechanical ventilation | 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Clara Vigneron, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin hospital, Paris, France, France

IPD SHARING:
Plan to Share IPD: No